CLINICAL TRIAL: NCT04863664
Title: Lead EvaluAtion for Defibrillation and Reliability (LEADR) / Lead Evaluation for Defibrillation and Reliability in Left Bundle Branch Area Pacing (LEADR LBBAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT19004 / MDT22048
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-04

CONDITIONS: Tachyarrhythmia
MeSH Terms: conditions — Tachycardia | interventions — Electric Countershock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Intervention/Treatment (LEADR) (Experimental): Patients will be implanted with a Next Generation ICD Lead and undergo required electrical testing
  Interventions: Device: Defibrillation (RV Implant)
- Intervention/Treatment (LEADR LBBAP) (Experimental): Patients will be implanted with a Next Generation ICD Lead in the LBBAP location and undergo required electrical testing
  Interventions: Device: Defibrillation (LBBAP Implant)

INTERVENTIONS:
Device: Defibrillation (RV Implant) — Required electrical testing for pacing, sensing, impedance and defibrillation will be completed
  Arms: Intervention/Treatment (LEADR)
Device: Defibrillation (LBBAP Implant) — Required electrical testing for pacing, sensing, impedance and defibrillation will be completed
  Arms: Intervention/Treatment (LEADR LBBAP)

SUMMARY:
The LEADR study is designed to assess the safety and efficacy of the Next Generation ICD lead.

The LEADR LBBAP study is being conducted under the existing US FDA Investigational Device Exemption (IDE) for the Next Generation ICD Lead and is designed to confirm the safety and defibrillation efficacy of the Next Generation ICD Lead when placed in the LBBAP location in ICD and LOT-CRT patient population.

DETAILED DESCRIPTION:
The LEADR and LEADR LBBAP studies will enroll subjects who are indicated to receive an implantable single or dual chamber ICD, or CRT-D, and who meet all of the inclusion criteria and none of the exclusion criteria. Subjects will receive an investigational Next Generation ICD Lead. Subjects in the LEADR study will be followed for at least 18 months following Next Generation ICD Lead implantation in a septal (non-LBBAP) or apical implant location. Enrollment in the LEADR study has been completed (675 subjects enrolled). Subjects in the LEADR LBBAP study will be followed for at least 3 months (ICD-indicated subjects) or 6 months (CRT-indicated subjects) following Next Generation ICD Lead implantation in an LBBAP implant location. Enrollment in the LEADR LBBAP study has been completed (323 subjects enrolled).

ELIGIBILITY:
LEADR Inclusion Criteria:

* Subject meets current clinical practice guidelines for implantation of ICD or CRT-D and will undergo one of the following:

  * de novo Medtronic CRT-D system implant
  * de novo Medtronic ICD system implant (single or dual chamber)
* Subject has, per local law and requirements, the minimum age for autonomously signing an ICF (minimum age of 18 years)
* Subject is willing to undergo implant defibrillation testing if requested.
* Subject is geographically stable and willing and able to complete the study procedures and visits for the duration of the follow-up.

LEADR Exclusion Criteria:

* Subject is unwilling or unable to personally provide Informed Consent.
* Subject has contraindications for standard RV transvenous lead placement (e.g., mechanical right heart valve).
* Subject is contraindicated for ≤1 mg dexamethasone acetate.
* Subject has a life expectancy of less than 12 months
* For subject undergoing defibrillation testing the following medical conditions exclude them:

  * Pre-existing or suspected pneumothorax during implant
  * Current intracardiac left atrial or left ventricular (LV) thrombus
  * Severe aortic stenosis
  * Severe proximal three-vessel or left main coronary artery disease without revascularization
  * Unstable angina
  * Ejection Fraction less than 25%
  * Recent stroke or transient ischemic attack (within the last 6 months)
  * Known inadequate external defibrillation
  * Any other known medical condition not listed that precludes their participation in the opinion of the investigator
* Subject is enrolled or planning to enroll in a concurrent clinical study that may confound the results of this study, without documented pre-approval from a Medtronic study manager.
* Subject with any exclusion criteria as required by local law (e.g., age or other).
* Pregnant women or breastfeeding women, or women of childbearing potential and who are not on a reliable form of birth regulation method or abstinence
* Subject with an existing pacemaker (including transcatheter pacing system), ICD, or CRT device or leads
* Subject with any evidence of active infection or undergoing treatment for an infection
* Recent (or planned) cardiac surgery or stenting less than 1 month before implant
* End stage renal disease
* Subjects with NYHA IV classification
* Subjects with a transplanted heart
* Subjects with previously extracted leads
* Subjects with Left Ventricular Assist Device

LEADR LBBAP Inclusion Criteria:

* Subject meets current local clinical practice guidelines for implantation of ICD (single or dual chamber) or CRT-D system and will undergo one of the following:

  a) De novo Medtronic ICD system implant (single or dual chamber) or b) De novo Medtronic CRT-D system implant and is intended to also undergo LV lead implant (for patients indicated for CRT-D according to locally approved indications/indications)
* Subject is 12 years of age or older and also is greater than 30 kg in weight at time of enrollment, has cardiac anatomy conducive to RV coil placement, and is allowed to participate in study per local law and requirements. Subjects from 12 years of age until adult also have a separate indication for pacing or CRT or are anticipated to develop one.
* Subject provides written authorization and/or consent per institution and geographical requirements.
* Subject is geographically stable and willing and able to complete the study procedures and visits for the duration of the follow-up
* Subject is willing to undergo implant defibrillation testing if requested

LEADR LBBAP Exclusion Criteria:

* Subject has contraindication for screw-in active fixation transvenous lead placement (e.g., mechanical right heart valve)
* Subject is contraindicated for ≤1 mg dexamethasone acetate
* Subject has a life expectancy of less than 12 months
* For subject undergoing defibrillation testing the following medical conditions exclude them:

  * Pre-existing or suspected pneumothorax
  * Current intracardiac left atrial or LV thrombus
  * Severe aortic stenosis
  * Severe proximal three-vessel or left main coronary artery disease without revascularization
  * Unstable angina
  * Recent stroke or transient ischemic attack (within the last 6 months)
  * Known inadequate external defibrillation
  * Any other known medical condition not listed that precludes their participation in the opinion of the investigator
* Subject is enrolled or planning to enroll in a concurrent clinical study that may confound the results of this study, without documented pre-approval from a Medtronic study manager
* Subject is pregnant or breastfeeding, or subject is of childbearing potential and not on a reliable form of birth regulation method or abstinence
* Subject with an existing pacemaker (including transvenous and transcatheter pacing system), ICD (transvenous) or CRT-D (transvenous) device or leads
* Subject with previous subcutaneous ICD (S-ICD), extravascular ICD (EV ICD) or Implantable Cardiac Monitor explanted within 30 days before implant
* Subject with any evidence of active bacterial infection or undergoing treatment for a bacterial infection within the last 30 days
* Recent (or planned) cardiovascular intervention within 30 days before or after implant, such as cardiac surgery, cardiac ablation, Percutaneous Coronary Intervention (PCI), or temporary cardiac pacing for >12 hours
* Subjects with end stage renal disease
* Subjects with NYHA IV classification
* Subjects with a transplanted heart or on the waiting list for a heart transplant
* Subjects with previously extracted leads
* Subjects with Left Ventricular Assist Device
* Subjects that are vulnerable adults

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 998 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
LEADR: Estimate the rate of major Lead complication-free rate at 6 months | Implant to 6 Months
  Subjects free of Next Generation ICD lead-related complication at 6 months post-implant.
LEADR: Percentage of subjects successfully defibrillated at implant with the Next Generation ICD lead | Day 1
  Defibrillation testing will be completed in a subset of subjects at implant.
LEADR LBBAP: Percentage of subjects successfully defibrillated at implant with the Next Generation ICD lead | Day 1
  Defibrillation testing will be completed with the Next Generation ICD Lead in the LBBAP location in a subset of subjects at implant.
LEADR LBBAP: The lead-related major complication rate at 3-months | Implant to 3 Months
  Subjects free of Next Generation ICD lead-related complication at 3 months post-implant.

SECONDARY OUTCOMES:
LEADR: Estimate the fracture-free rate of the Next Generation ICD lead | up to 24 months
  Subjects will be assessed at certain time points for Next Generation ICD lead fracture related to the Next Generation ICD lead.

CONTACTS AND LOCATIONS:
Overall Officials: George Crossley, MD, Principal Investigator — Vanderbilt University (LEADR); Pugazhendhi Vijayaraman, MD, Principal Investigator — Geisinger Medical Center (LEADR LBBAP)
Locations (55):
- United States (23):
  - LEADR: Heart Center Research, Huntsville, Alabama
  - LEADR LBBAP: Torrance Memorial Medical Center, Torrance, California
  - LEADR: Hartford Hospital, Hartford, Connecticut
  - LEADR: University of South Florida, Tampa, Florida
  - LEADR & LEADR LBBAP: Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - LEADR: Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - LEADR: Washington University School of Medicine, St Louis, Missouri
  - LEADR: Lourdes Cardiology Services, Voorhees Township, New Jersey
  - LEADR: Presbyterian Heart Group, Albuquerque, New Mexico
  - LEADR & LEADR LBBAP: South Shore University Hospital/Northwell Health, Bay Shore, New York
  - LEADR: TriHealth Hatton Research Institute, Cincinnati, Ohio
  - LEADR LBBAP: The Christ Hospital, Cincinnati, Ohio
  - LEADR: Cleveland Clinic, Cleveland, Ohio
  - LEADR LBBAP: The Ohio State University Wexner Medical Center, Columbus, Ohio
  - LEADR: Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - LEADR: Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - LEADR LBBAP: Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - LEADR& LEADR LBBAP: Vanderbilt University medical Center, Nashville, Tennessee
  - LEADR: Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - LEADR: Texas Health Fort Worth Hospital, Fort Worth, Texas
  - LEADR & LEADR LBBAP: University of Virginia Medical Center, Charlottesville, Virginia
  - LEADR & LEADR LBBAP: Virginia Commonwealth University Health System, Richmond, Virginia
  - LEADR LBBAP: Aurora St. Luke's Hospital, Milwaukee, Wisconsin
- Australia (4):
  - LEADR & LEADR LBBAP: The Prince Charles Hospital, Chermside, Queensland
  - LEADR: Ashford Hospital, Ashford, South Australia
  - LEADR & LEADR LBBAP: Royal Adelaide, Norwood, South Australia
  - LEADR &LEADR LBBAP: Canberra Hospital, Garran
- LEADR: Universitätsklinikum Krems, Krems, Mitterweg, Austria
- LEADR LBBAP: Universitair Ziekenhuis Antwerpen, Edegem, Antwerp, Belgium
- Canada (3):
  - LEADR: University of Calgary, Calgary, Alberta
  - LEADR: Southlake Regional Health Centre, Newmarket, Ontario
  - LEADR & LEADR LBBAP: Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
- China (2):
  - LEADR: Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - LEADR & LEADR LBBAP: West China Hospital of Sichuan University, Chengdu
- LEADR: Rigshospitalet, Copenhagen, Denmark
- France (3):
  - LEADR: Centre Hospitalier Universitaire de Grenoble - Site Nord, La Tronche
  - LEADR LBBAP: OC Santé - Clinique du Millénaire, Montpellier
  - LEADR: CHU Hôpitaux de Rouen - Hôpital Charles Nicolle, Rouen
- LEADR: Klinikum Bielefeld Kardiologie, Bielefeld, Bielefeld, Germany
- Hong Kong (2):
  - LEADR & LEADR LBBAP: Queen Mary Hospital, Hong Kong
  - LEADR: Princess Margaret Hospital, Lai Chi Kok
- LEADR: Azienda Socio Sanitaria Territoriale (ASST) Papa Giovanni XXIII, Bergamo, Italy
- Japan (3):
  - LEADR & LEADR LBBAP: Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - LEADR & LEADR LBBAP: National Cerebral and Cardiovascular Center, Suita, Osaka
  - LEADR: Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo
- LEADR & LEADR LBBAP: Institut Jantung Negara - National Heart Institute, Kuala Lumpur, Malaysia
- LEADR LBBAP: Maastricht Universitair Medisch Centrum, Maastricht, Limburg, Netherlands
- LEADR LBBAP: Szpital Uniwersytecki w Krakowie, Krakow, Poland
- LEADR: Centro Hospitalar de Lisboa Ocidental, E.P.E. Hospital de Santa Cruz Cardiology, Carnaxide, Portugal
- LEADR: Klinicki Centar Srbije Pejsmejker centar, Belgrade, Serbia
- LEADR: Ng Teng Fong General Hospital, Singapore, Singapore, Singapore
- Spain (3):
  - LEADR LBBAP: Hospital Universitario Virgen de las Nieves, Granada, Granada
  - LEADR: Hospital Universitari Bellvitge, L'Hospitalet de Llobregat
  - LEADR: Hospital Universitario y Politécnico La Fe, Valencia
- LEADR & LEADR LBBAP: Imperial College Healthcare NHS Trust - Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crossley GH 3rd, Mason PK, Hansky B, De Filippo P, Shah MJ, Philippon F, Sholevar D, Richardson TD, West MB, Dinerman J, Dawson J, Himes A, Severseike L, Thompson AE, Sanders P. High predicted durability for the novel small-diameter OmniaSecure defibrillation lead. Heart Rhythm. 2025 Feb;22(2):302-310. doi: 10.1016/j.hrthm.2024.09.005. Epub 2024 Sep 26. PMID 39341436